CLINICAL TRIAL: NCT06601348
Title: Effectiveness of a School-Based Nutrition Education and Physical Activity Intervention for Overweight and Obese Children: the Health Promoting School (Hps) Model
Brief Title: The Effectiveness of the Health Promoting School Intervention Model in Reducing Overweight and Obesity Among School Children in Indonesia: a Mixed-Methods Protocol Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Rosdiana, Effectiveness Of A School-Based Nutrition Education And Physical Activity Intervention For Overweight And Obese Children: The Health Promoting School (Hps) Model, Gadjah Mada University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KE/FK/1235/EC/2024
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Overweight and Obese Children
Keywords: Childhood overweight and obesity, health promoting schools, Nutrition Education, Physical activity
MeSH Terms: conditions — Overweight; Pediatric Obesity; Obesity; Motor Activity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nutrition education, physical activity interventions, and a health promoting school (Other): The intervention programme will be implemented for 6 months. Nutrition education is developed through piloting a health promoting school model, the content will combine the government programme "healthy school" and WHO cartoon pamphlets distributed to each school/student in the intervention school. Nutrition and health education was provided 6 times for students, and 2 times for parents and 4 times for teachers and UKS officers. Physical activity intervention School-based physical activity programme for students called "Happy in school children" Other forms of physical activity included games, dance or rhythmic gymnastics, such as jumping rope, and squatting, or by adjusting the curriculum. And piloting the health promoting school (HPS) model, the expected outcome of the health promoting school (HPS) model is health literacy.
  Interventions: Other: Nutrition education, physical activity intervention, and health promoting school model trials

INTERVENTIONS:
Other: Nutrition education, physical activity intervention, and health promoting school model trials — A nutrition education and physical activity intervention, combining a pilot health promoting school model that includes health education and recreational enhancement with the curriculum of a government-designated healthy school, was designed to reduce childhood overweight and obesity. The programme was implemented over 6 months. This program has been widely conducted in several countries, but there are still many differences from previous studies, especially in terms of strengthening qualitative studies in the first stage, then in the intervention stage using a Cluster Randomised Controlled Trial design. Another advantage of this study is the combination of intervention and health promoting school. In Indonesia, there are few intervention studies in reducing overweight and obesity in children, some only focus on descriptive studies such as nutritional knowledge, physical activity measures using questionnaires to determine the relationship or measure BMI.

SUMMARY:
The prevalence of obesity in children is increasing rapidly, Among children aged 5-12 years, 18.8% have severe overweight, comprising 10.8% who are obese and 8.8% who are over. The development of effective and sustainable intervention strategies to prevent childhood obesity in Indonesia is becoming increasingly important, particularly given the limited implementation of health-promoting schools in the country.

The first Phase using qualitative exploration was a needs assessment will be using of social cognitive theory. The second Phase will be the development model intervention modification of the health promotion school WHO and "Health School". The third Phase is the quantitative stage using a Cluster Randomised Controlled Trial to analyse differences and test the effectiveness of the HPS model. This study will be conducted in 8 primary schools located in Makassar, South Sulawesi. School in Makassar city and schools from outside Makassar city, randomly selected for the trial. Then the selected schools are randomly divided into school for nutrition education and physical activity. Intervention, while school each for comprehensive intervention. The study will be target students in Grades 4 and 5 of primary school. Assessments for the primary objective (BMI Z score), and secondary objectives (change in knowledge, self-efficacy, and health literacy) in thirds study arm. The subsequent phase will assess the efficacy of the intervention in terms of reductions in BMI Z scores, improvements in knowledge, self-efficacy and health literacy. Concurrently, the exploration of parental and teacher knowledge and insights regarding health promotion in schools and its potential in reducing overweight and obesity in children will be conducted.

DETAILED DESCRIPTION:
This research is an exploratory sequential mixed method design. By combining two elements of qualitative and quantitative research approaches. Exploratory sequential mixed method. The qualitative phase includes an exploration of needs assessment with a social cognitive theory approach, the second phase implements the Health Promoting School model for three months. The third phase was quantitative using Cluster Randomised Controlled Trial design. To analyse the effectiveness of a 6-month school-based intervention in children aged 9 and 12 years in schools with A and B accreditation standards. Three interventions will be implemented and outcomes will be measured simultaneously. Sampling in the study, using two steps in the selection of subjects, first 8 schools from the city of Makassar and 4 schools outside the city of Makassar from each school were randomly selected for the trial. then the selected schools were randomly divided into 4 groups, for nutrition education and physical activity interventions, while 4 groups each for comprehensive interventions. Inclusion criteria for selecting schools: 1) non- boarding schools; 2) the prevalence of obesity, based on routine physical examination records, was above 10%; 3) school lunch was provided, and more than 50% of students ate school lunch. All students in the selected classes were invited to participate in the study.

Exclusion criteria for subjects: 1) students suffering from serious diseases (such as congenital heart disease, or other diseases and so on) or unable to withstand strenuous physical activity or dietary regulation were excluded. 2) Students participating in the study or intending to transfer to another similar school in the following year are excluded.

This study will be conducted in Makassar, Gowa and Maros cities in South Sulawesi. The unit of analysis for this study is primary schools, especially in Makassar and other cities. A preliminary study was conducted at all school sites to determine the number of students who would fit the special criteria of 9-12 years of age in primary school children at eight schools in South Sulawesi who were willing to participate in the study. There were eight schools in this study that met these criteria SDN Athira, SD Al-Ashar, SDN Pallangga Gowa, SD Sudirman, SD Alfityan, SDN Tete Batu 1 SDN Tete Batu, and SDN Bulurokeng. The results of the preliminary study showed that the number of overweight and obese students at SDN Athira was 39.4%, SDN Pallangga 27.5%, SD Sudirmana I 45.5%, SD Tete Batu 49.7%, SD Alashar 26.2%, and SD Alfityan 58.7%, SDN Tete Batu I 50.8%, and SDN Bulurokeng 45.7%. Furthermore, from these eight primary schools, the primary schools that will be given the intervention and their willingness to continue their participation in the intervention and implementation of the HPS model for reducing overweight and obesity in primary school children were selected. Based on these criteria, these are the primary schools that will be treated.

Student recruitment: all grade 4 and 5 students who met the inclusion criteria were verbally informed about the study at the time of recruitment. Written information will be given to parents or guardians for them to study and ask them to give informed consent if they agree to their child taking part in the study. Recruitment of UKS teachers, science and sports teachers, or homeroom teachers: with permission from the principals of primary schools willing to participate in the study.

The sample size in this study was determined based on the formula for hypothesis testing of mean differences between intervention. The calculation uses the formula as follows :

All data were presented as mean (SD) or median, range, or percentage (for categorical variations). Statistics analyzed will be used software SPSS and STATA. The normality test used the Shapiro-Wilk test. At baseline measurement, anova test was performed to determine the difference between effectivites. After follow-up, within-group were compared by independent t-test. Comparison of before and after variables was assessed wiil be paired t- test for normally distributed data, or by Mann-Whitney test for non-normally distributed data was considered statistic significant if the P- value of less thsn 0.05 will be considered statiscally. Effect size will be measured using Cohen d. To see the comparison of outcomes measured in months two, four and six will be tested using repeated annova. Analysis of covariance (ANCOVA) was used to test the outcomes that have an effect on the effectiveness of the HPS model and nutrition education and physical activity interventions in overweight and obese children.

Analysis qualitatif with transcripts from all focus groups will be independently analysed by two researchers will be using thematic analysis. The thematic analysis will consist of a six-step approach which includes; (i) data familiarisation achieved by reading each transcript, (ii) initial code generation, (iii) theme search from initial codes, (iv) thematic map generation, (v) specific definition and naming of themes and (vi) final analysis. The two sets of thematic analyses will be compared before the final iteration of thematic analysis is conducted and final themes are generated and consensus is reached. Qualitative data contextual the results and investigates participants, perceptions and attitudes towards the intervention Data collection is done by giving pretest and posttest questionnaires to all children in the intervention group. At the time of data collection, students will be divided into groups. Each group of five students will be guided by an interviewer or facilitator when completing the questionnaire. Each student had to answer all the questions on the questionnaire on the same day. The head of the class emphasised to the students to fill in the questionnaire honestly and that the result of the questionnaire would not affect their rapport score. This is to obtain accurate data. In addition to filling out the questionnaire, anthropometric measurements were also taken on students by trained enumerators. These measurements will be taken on different days during designated hours and will be taken monthly for six months, in all groups.

ELIGIBILITY:
Inclusion Criteria:

* Male and female gender
* Children aged 9-12 years old (at the time of baseline data collection)
* All fourth and fifth grade students/children
* Children who are willing as respondents and ready to follow the intervention until completion and willing to fill in the informed consent.
* Withdrawal: Children experiencing physical and mental health conditions during the intervention (arising due to the child's own health conditions, not due to the effects of the intervention)
* Full day children

Exclusion Criteria:

* Children with clinical conditions / health disorders such as heart disease etc.)
* Children who did not take the pretest
* Children who left or moved schools
* Children who did not complete the intervention

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2024-10-04 (Estimated); Primary Completion 2025-05-18 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
BMI Z-score | 6 months intervention combining health promoting school
  Where weight will be measured using a body composition meter (Seca 804) to 0.1 kg, and height measured with a stadiometer to 0.1 cm. BMI (kg/m2) will be converted to the Weight and height measurements will be taken twice to obtain accuracy and correct averages. Body mass index (BMI) for age Z score, according in 2007 WHO Growth Standards for children, will be used to classify the risk of being overweight with a Z SD score of 1, overweight with a Z SD score 1, and overweight: BMI Z-score ≤ 3, obesity BMI Z- score ≥ 3.

SECONDARY OUTCOMES:
Children knowledge, Self-efficacy, and Health Literacy | 3 months trial, 3 months implementation of health promoting school (HPS) model
  Children knowledge, the ability to give appropriate answers to questions about nutrition, physical activity, causes of overweight and obesity and how to prevent them. The measuring instrument uses a questionnaire, a ratio measuring scale, the measurement result is determined from the total score set, the correct answer score is given 1) if it is wrong 0).
  Self-efficacy, a person belief in their ability to perform a behaviour, the behaviour is obesity prevention, measured using a 3-point Likert scale, namely 1) agree, 2) disagree, and 3) disagree. Answer score for favourable questions: Agree: 3) Undecided: 2) Disagree:1) Unfavourable question answer score: Agree: 1) Undecided: 2) Disagree: 3).
  Health literacy, the ability of children, orangutans and schools to apply and use information, health promoting school approach measurement tool, in-depth interview and questionnaire distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Toto Sudargo, Ph.D, Study Director — Gadjah Mada University
Locations (2):
- Indonesia (2):
  - Elementary School Al-Azhar, Makassar, South Sulawesi
  - Elementary School Tete Batu and Sudirman, Makassar, South Sulawesi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Z, Xu F, Ye Q, Tse LA, Xue H, Tan Z, Leslie E, Owen N, Wang Y. Childhood obesity prevention through a community-based cluster randomized controlled physical activity intervention among schools in china: the health legacy project of the 2nd world summer youth olympic Games (YOG-Obesity study). Int J Obes (Lond). 2018 Apr;42(4):625-633. doi: 10.1038/ijo.2017.243. Epub 2017 Oct 5. PMID 28978975
- [Background] Pluimakers VG, van Atteveld JE, de Winter DTC, Bolier M, Fiocco M, Nievelstein RJAJ, Janssens GOR, Bresters D, van der Heiden-van der Loo M, de Vries ACH, Louwerens M, van der Pal HJ, Pluijm SMF, Ronckers CM, Versluijs AB, Kremer LCM, Loonen JJ, van Dulmen-den Broeder E, Tissing WJE, van Santen HM, van den Heuvel-Eibrink MM, Neggers SJCMM. Prevalence, risk factors, and optimal way to determine overweight, obesity, and morbid obesity in the first Dutch cohort of 2338 long-term survivors of childhood cancer: a DCCSS-LATER study. Eur J Endocrinol. 2023 Nov 8;189(5):495-507. doi: 10.1093/ejendo/lvad139. PMID 37837608
- [Background] Lee J, Hoornbeek J, Oh N. Social Cognitive Orientations, Social Support, and Physical Activity among at-Risk Urban Children: Insights from a Structural Equation Model. Int J Environ Res Public Health. 2020 Sep 16;17(18):6745. doi: 10.3390/ijerph17186745. PMID 32947944
- [Background] Caballero B, Clay T, Davis SM, Ethelbah B, Rock BH, Lohman T, Norman J, Story M, Stone EJ, Stephenson L, Stevens J; Pathways Study Research Group. Pathways: a school-based, randomized controlled trial for the prevention of obesity in American Indian schoolchildren. Am J Clin Nutr. 2003 Nov;78(5):1030-8. doi: 10.1093/ajcn/78.5.1030. PMID 14594792
- [Background] Almutairi N, Burns S, Portsmouth L. Barriers and enablers to the implementation of school-based obesity prevention strategies in Jeddah, KSA. Int J Qual Stud Health Well-being. 2022 Dec;17(1):2135197. doi: 10.1080/17482631.2022.2135197. PMID 36263729
- [Background] Bartelink NHM, van Assema P, Kremers SPJ, Savelberg HHCM, Oosterhoff M, Willeboordse M, van Schayck OCP, Winkens B, Jansen MWJ. Can the Healthy Primary School of the Future offer perspective in the ongoing obesity epidemic in young children? A Dutch quasi-experimental study. BMJ Open. 2019 Oct 31;9(10):e030676. doi: 10.1136/bmjopen-2019-030676. PMID 31676651
- See also: Related Info — https://bmjopen.bmj.com/content/9/10/e030676
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9590444/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32947944/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37837608/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28978975/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/14594792/